CLINICAL TRIAL: NCT00244153
Title: Intraarticular Application of Opioids Versus Glucocorticosteroids Versus Placebo in Rheumatoid Arthritis
Brief Title: Intraarticular Opioids Vs Glucocorticosteroids in Gonarthritis
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Mor01
Record Dates: First submitted 2005-10-25; First posted 2005-10-26 (Estimated); Last update posted 2006-09-11 (Estimated); Status verified 2004-02

CONDITIONS: Rheumatic Disease
Keywords: intraarticular morphine, steroids, arthroscopy
MeSH Terms: conditions — Rheumatic Diseases

INTERVENTIONS:
Drug: intraarticular morphine
Drug: intraarticular dexamethasone

SUMMARY:
Intraarticular application of opioids versus glucocorticosteroids versus placebo in knee arthritis

study goals: assessment of effectiveness and tolerability of locally applied morphine, dexamethasone or placebo in knee arthritis

DETAILED DESCRIPTION:
Study background

Patients with chronic inflammatory arthritis (e.g. rheumatoid arthritis, undifferentiated oligoarthritis, monarthritis) suffer from recurrent pain, functional impairment and impaired capacity. Consequences of such hard to treat diseases are occupational incapacity and early retirement. The treatment options we have today such as nonsteroidal antirheumatic drugs (NSAIDs such as diclofenac), glucocorticosteroids (e.g. dexamethasone) and disease modifying antirheumatic drugs (such as methotrexate) partly are effective but also have serious side effects and complications (e.g. gastric and duodenal ulcers, nephrotoxicity, degeneration of cartilage, cushing´s syndrome…).

A new therapeutic approach without such complications is represented by the intraarticular (i.a.) application of low-concentrated, systemically inactive dosages of an opioid (e.g. morphine). This treatment showed a significant reduction of pain in patients with chronic arthritis in controlled clinical trials without systemic or local side effects [1, 2]. This effect is based on an activation of peripheral opioid receptors, which could be identified on peripheral nerve endings of sensoric neurons [3-5]. The activation of these opioid receptors leads to a decrease of neuronal excitability and the transmission of noziceptive impulses as well as to a reduced release of proinflammatory neurotransmitters (e.g. substance p) [6]. Several studies showed that locally applied opioids act analgetic, that such analgetic effects mainly occur in inflamed tissue, that the analgetic effects increase with the degree of inflammation and that peripherally acting opioids act analgetic [6-9]. In human beings the analgetic effect of peripherally applied opioid agonists has almost only been shown in patients with acute post-surgical pain [4, 10-15]. In a first case report [16] we found indices for the analgetic effect of i.a. given morphine in patients with chronic arthritic pain. In patients with osteoarthritis a double blind cross-over study it was shown that 1mg morphine leads to a long-lasting analgetic effect up to 9 days [1]. In a second controlled trial we compared patients with chronic joint inflammation in different diseases in regards of the analgetic effect of i.a. morphine (3 mg) versus placebo versus a standard therapy with i.a. dexamethasone (4 mg) [2]. Dexamethasone as well as morphine lead to a significant pain reduction under rest and under strain compared to placebo. This analgetic effect lasted up to 6 days after injection. Moreover we found first indications for an anti-inflammatory effect as the number of inflammatory cells in the synovial fluid was reduced after the i.a. morphine application [2].

In addition to the question whether morphine can stimulate local peripheral opioid receptors, it should be investigated, whether intraarticular morphine has an anti-inflammatory local effect in arthritis of the knee in the setting of inflammatory rheumatic diseases such as rheumatoid arthritis, spondyloarthropathies, undifferentiated oligoarthritis or monarthritis (17, 19, 31). This question should be answered through investigation of cellular infiltration and cytokine expression in the synovial membrane and synovial fluid.

Next to the exogenous application of opioids also endogenous opioid peptides play an important role in inflammatory processes. Experimental and clinical investigations show an expression of opioid peptides in immune cells, which invade into inflamed tissue [3, 4, 6, 20, 21]. Under certain circumstances these opioid peptides are locally released and unfold a strong analgetic effect through the activation of opioid receptors on peripheral sensoric nerve endings [22-24]. Corticotropin-releasing factor (CRF) can release - similar as in the hypophysis- opioid peptides from immune cells [25-28]. CRF receptors are located in regionally invaded immune cells, and the number is up regulated among inflammatory cells. [29]. Experimental investigations from our or other groups showed a significant analgetic effect of local CRF which was given into the inflamed tissue [24, 26, 30].

In this study we want to test the hypothesis, that i.a. applied CRF leads to a reduction of pain intensity and pain duration in patients with inflammatory knee trauma. Initially this effect is to be tested in acute and then - if successful- in chronic knee pain.

Background for dosage

The intraarticular application of morphine 3mg and dexamethasone 4 mg respectively has turned out from previous studies (2, 15) in patients with inflammatory knee joints of different causes, without evidence of relevant systemic side effects.

Background for patient selection:

Several patients with inflammatory rheumatic diseases such as rheumatoid arthritis, spondyloarthropathies, undifferentiated oligoarthritis or monarthritis suffer from symptomatic knee arthritis despite intake of disease modifying drugs (DMARDs) or systemic low dose glucocorticosteroids. To achieve a adequate comparability of the different drugs a patient number of 20 for each group seems to be sufficient. Patients are supposed to have arthritis of the knee and a sufficient pain intensity according to the visual analogue scale for pain > 30 mm. Patients will be seen in the rheumatology department of the Klinikum Benjamin-Franklin, Berlin, Germany as well as in the Immanuel-Krankenhaus, Berlin, Germany examined. Arthroscopies will only take place in the rheumatology department of the Klinikum Benjamin-Franklin, Berlin, Germany.

References:

1. Likar R, Schäfer M, Paulak F, et al. Intraarticular morphine analgesia in chronic pain patients with osteoarthritis. Anesth Analg 1997;84:1313-7.
2. Stein A, Yassouridis A, Szopko C, Helmke K, Stein C. Intraarticular morphine versus dexamethasone in chronic arthritis. Pain 1999;83:525-32.
3. Stein C. The control of pain in peripheral tissue by opioids. N Engl J Med 1995;332:1685-90.
4. Stein C, Pflüger M, Yassouridis A, et al. No tolerance to peripheral morphine analgesia in presence of opioid expression in inflamed synovia. J Clin Invest 1996;98:793-9.
5. Mousa SA, Zhang Q, Sitte N, Ji R, Stein C. beta-Endorphin-containing memory-cells and mu-opioid receptors undergo transport to peripheral inflamed tissue. J Neuroimmunol 2001;115:71-8.
6. Stein C, Machelska H, Schäfer M. Peripheral analgesic and antiinflammatory effects of opioids. Z Rheumatol 2001;60:416-24.
7. Binder W, Walker JS. Effect of the peripherally selective kappa-opioid agonist, asimadoline, on adjuvant arthritis. Br J Pharmacol 1998;124:647-54.
8. Wilson JL, Walker JS, Antoon JS, Perry MA. Intercellular adhesion molecule-1 expression in adjuvant arthritis in rats: inhibition by kappa-opioid agonist but not by NSAID. J Rheumatol 1998;25:499-505.
9. Binder W, Machelska H, Mousa S, et al. Analgesic and antiinflammatory effects of two novel kappa opioid peptides. Anesthesiology 2001;94:1034-44.
10. Stein C, Comisel K, Haimerl E, et al. Analgesic effect of intraarticular morphine after arthroscopic knee surgery. N Engl J Med 1991;325:1123-6.
11. Khoury GF, Chen ACN, Garland DE, Stein C. Intraarticular morphine, bupivacaine and morphine/bupivacaine for pain control after knee videoarthroscopy. Anesthesiology 1992;77:263-6.
12. Likar R, Kapral S, Steinkellner H, Stein C, Schäfer M. Dose-dependency of intra-articular morphine analgesia. Br J Anaesth 1999;83:241-4.
13. Schäfer M. Peripheral opioid analgesia: from experimental to clinical studies. Curr Opin Anaesth 1999;12:603-7.
14. Gupta A, Bodin L, Holmstrom B, Berggren L. A systematic review of the peripheral analgesic effects of intraarticular morphine. Anesth Analg 2001;93:761-70.
15. Kalso E, Smith L, McQuay HJ, Moore A. No pain, no gain: clinical excellence and scientific rigour - lessons learned from IA morphine. Pain 2002;98: 269-275.
16. Khoury GF, Garland DE, Stein C. Intraarticular opioid-local anesthetic combinations for chronic joint pain. Middle East J Anesth 1994;12:579-85.
17. Simon AK, Seipelt E, Sieper J. Divergent T-cell cytokine patterns in inflammatory arthritis. Proc Natl Acad Sci U S A 1994;91:8562-6.
18. Yin Z, Siegert S, Neure L, et al. The elevated ratio of interferon gamma-/interleukin-4-positive T cells found in synovial fluid and synovial membrane of rheumatoid arthritis patients can be changed by interleukin-4 but not by interleukin-10 or transforming growth factor beta. Rheumatology (Oxford) 1999;38:1058-67.
19. Rudwaleit M, Yin Z, Siegert S, et al. Response to methotrexate in early rheumatoid arthritis is associated with a decrease of T cell derived tumour necrosis factor alpha, increase of interleukin 10, and predicted by the initial concentration of interleukin 4. Ann Rheum Dis 2000;59:311-4.
20. Machelska H, Cabot PJ, Mousa SA, Zhang Q, Stein C. Pain control in inflammation governed by selectins. Nature Med 1998;4:1425-8.
21. Rittner HL, Brack A, Machelska H, et al. Opioid peptide-expressing leukocytes: identification, recruitment, and simultaneously increasing inhibition of inflammatory pain. Anesthesiology 2001;95:500-8.
22. Stein C, Hassan AHS, Przewlocki R, Gramsch C, Peter K, Herz A. Opioids from immunocytes interact with receptors on sensory nerves to inhibit nociception in inflammation. Proc Natl Acad Sci USA 1990;87:5935-9.
23. Stein C, Hassan AHS, Lehrberger K, Giefing J, Yassouridis A. Local analgesic effect of endogenous opioid peptides. Lancet 1993;342:321-4.
24. Schäfer M, Carter L, Stein C. Interleukin-1 and corticotropin-releasing-factor inhibit pain by releasing opioids from immune cells in inflamed tissue. Proc Natl Acad Sci USA 1994;91:4219-23.
25. Schäfer M, Mousa SA, Zhang Q, Carter L, Stein C. Expression of corticotropin-releasing factor in inflamed tissue is required for intrinsic peripheral opioid analgesia. Proc Natl Acad Sci USA 1996;93:6096-100.
26. Lariviere WR, Melzack R. The role of corticotropin-releasing factor in pain and analgesia. Pain 2000;84:1-12.
27. Cabot PJ, Carter L, Gaiddon C, et al. Immune cell-derived -endorphin: production, release and control of inflammatory pain in rats. J Clin Invest 1997;100:142-8.
28. Cabot PJ, Carter L, Schäfer M, Stein C. Methionine-enkephalin- and Dynorphin A-release from immune cells and control of inflammatory pain. Pain 2001;93:207-12.
29. Mousa SA, Schäfer M, Mitchell WM, Hassan AHS, Stein C. Local upregulation of corticotropin- releasing hormone and interleukin-1 receptors in rats with painful hindlimb inflammation. Eur J Pharmacol 1996;311:221-31.
30. Schäfer M, Mousa SA, Stein C. Corticotropin-releasing factor in antinociception and inflammation. Eur J Pharmacol 1997;323:1-10.
31. Leirisalo-Repo M. Prognosis, course of disease, and treatment of the spondyloarthropathies. Rheum Dis Clin North Am. 1998 Nov;24(4):737-51

ELIGIBILITY:
Inclusion Criteria:

* Arthritis according to the American Rheumatism Association or osteoarthritis of the knee
* age older than 18 years
* active gonarthritis in the setting of a rheumatic inflammatory disease such as rheumatoid arthritis, spondyloarthropathies, undifferentiated oligoarthritis or monarthritis since at least 4 weeks with proof of joint or ostearthritis of the knee effusion in ultrasound
* visual analogue scale (pain) >30 mm
* weight between 50 and 90 kg
* signed informed consent
* negative urine pregnancy test in women of child-bearing potential

Exclusion Criteria:

* pregnancy / lactation
* severe infection, suspicion for opportunistic infection within the last 2 months (herpes zoster, cytomegaly-, pneumocystis carinii-infection), HIV- infection
* malignant disease
* severe cardiac, renal, hematologic, pulmonary, neurologic, gastrointestinal (amongst others gastric or duodenal ulcer) or hepatic (viral hepatitis, toxic liver disease etc) disease, uncontrolled high blood pressure, recurrent thrombosis/ embolism
* psychiatric disease
* significant bone marrow dysfunction with impaired hematopoiesis
* one of the following laboratory findings: thrombocytopenia < 100 /nl, Quick < 50%
* significant pathological findings in physical examination, especially findings indicating an infectious cause for arthritis (septic arthritis) or Lyme arthritis
* participation in clinical trials within the last 30 days
* intake of illegal drugs (such as cocaine, heroin...), substance abuse (alcohol, excessive intake of analgetic drugs, benzodiazepines)
* intake of anticoagulating drugs

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120
Dates: Start 2004-06; Study Completion 2007-08

PRIMARY OUTCOMES:
primary endpoints: improvement on the visual analogue scale (VAS) of minimally 20mm on a scale from 0- 100mm

SECONDARY OUTCOMES:
secondary end points: improvement of the numeric rating scale, quality of sleep, global daily activity, WOMAC, improvement of joint mobility according to the Lysholm and Gillquist scores and improvement of pain on a four digit scale.

CONTACTS AND LOCATIONS:
Overall Officials: Joachim Sieper, Prof., Principal Investigator — Charité Campus Benjamin-Franklin, Rheumatology
Locations (1):
- Immanuel Krankenhaus, Berlin, Germany